CLINICAL TRIAL: NCT00674206
Title: A Phase II Trial of Gemcitabine and Oxaliplatin for ER-, PR-, HER2NEU- (Triple Negative) Metastatic Breast Cancer
Brief Title: A Phase II Trial of Gemcitabine and Oxaliplatin for Triple Negative Metastatic Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor funding stopped
Sponsor: Emory University (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Principal Investigator, Amelia Zelnak, MD, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00007792; 7792 (Other: Other)
Record Dates: First submitted 2008-05-06; First posted 2008-05-07 (Estimated); Results first posted 2012-07-26 (Estimated); Last update posted 2013-12-12 (Estimated); Status verified 2013-11

CONDITIONS: Breast Cancer
Keywords: Metastatic breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Gemcitabine; gemcitabine-oxaliplatin regimen; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Gemcitabine and Oxaliplatin (Experimental): All patients enrolled on clinical trial will receive Gemcitabine 1000mg/m^2 on Day 1 and Oxaliplatin 100 mg/m^2 intravenously over 2 hours on Day 2.
  Interventions: Drug: Gemcitabine; Drug: Oxaliplatin

INTERVENTIONS:
Drug: Gemcitabine — Gemcitabine 1000mg/m^2 on day 1 every 14 days Cycles of treatment will be repeated every 2 weeks until disease progression, intolerable toxicity, or the development of any of the criteria for study removal
  Other Names: Gemcitabine, Oxaliplatin
Drug: Oxaliplatin — Oxaliplatin 100mg/m^2 on day 2 every 14 days Cycles of treatment will be repeated every 2 weeks until disease progression, intolerable toxicity, or the development of any of the criteria for study removal

SUMMARY:
The purpose of this study is to investigate if the combination of gemcitabine and oxaliplatin is effective for triple negative breast cancer.

DETAILED DESCRIPTION:
In this study, participants will receive gemcitabine and oxaliplatin, drugs that have been in use for a long time. Gemcitabine is a treatment that is an effective therapy currently available to patients with this type and stage of breast cancer. Frequently, in cancer therapy, combinations of drugs prove more effective as treatment than the same drugs used alone. The combination of gemcitabine and oxaliplatin has not been tested in patients with triple negative breast cancer. It is hoped that the addition of oxaliplatin may cause your tumor to stop growing or possible your tumor may shrink. This assessment will be basd on measuring changes in the size of your tumor.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed ER-, PR-, Her2neu- (Triple Negative) metastatic breast cancer
* Patients must have measurable disease according to the RECIST criteria. Patients with bone metastases may be included if they have a decrease in performance status or narcotic analgesic requirement.
* Patients must have either received a taxane in the adjuvant setting or received a taxane as first-line treatment for metastatic breast cancer
* Age > 18 years
* ECOG Performance Score of 0, 1, or 2 (Appendix A)
* Adequate bone marrow as evidenced by:
* Absolute neutrophil count > 1,500/L
* Platelet count > 100,000/microL
* Adequate renal function as evidenced by serum creatinine < 1.5 mg/dL
* Adequate hepatic function as evidenced by:

  * Serum total bilirubin < 1.5 mg/dL
  * Alkaline phosphatase < 3X the ULN for the reference lab < 5X the ULN (Upper limit for normal) for patients with known hepatic metastases
  * SGOT/SGPT < 3X the ULN(Upper limit for normal) for the reference lab (< 5X the ULN for patients with known hepatic metastases
* Patients must be recovered from both acute and late effects of any prior surgery, radiotherapy or other antineoplastic therapy
* Patients or their legal representatives must be able to read, understand and provide informed consent to participate in the trial.
* Patients of childbearing potential agree to use an effective form of contraception during the study and for 90 days following the last dose of study medication (an effective form of contraception is an oral contraceptive or a double barrier method)

Exclusion Criteria:

* Patients with an active infection or with a fever > 101.30 F within 3 days of the first scheduled day of protocol treatment
* Patients with active CNS metastases. Patients with stable CNS disease, who have undergone radiotherapy at least 4 weeks prior to the planned first protocol treatment and who have been on a stable dose of corticosteroids for 3 weeks are eligible for the trial
* History of prior malignancy within the past 5 years except for curatively treated basal cell carcinoma of the skin, cervical intra-epithelial neoplasia, or localized prostate cancer with a current PSA of < 1.0 mg/dL on 2 successive evaluations at least 3 months apart, with the most recent evaluation within 4 weeks of entry
* Patients with known hypersensitivity to any of the components of oxaliplatin or gemcitabine.
* Patients who have received gemcitabine or platin-based chemotherapy in the past.
* Patients who have received chemotherapy within 28 days of the first scheduled day of protocol treatment.
* Patients who received radiotherapy to more than 25% of their bone marrow; or patients who received any radiotherapy within 4 weeks of entry
* Patients who are receiving concurrent investigational therapy or who have received investigational therapy within 28 days of the first scheduled day of protocol treatment (investigational therapy is defined as treatment for which there is currently no regulatory authority approved indication)
* Peripheral neuropathy Grade 2
* Patients who are pregnant or lactating
* Any other medical condition, including mental illness or substance abuse, deemed by the Investigator to be likely to interfere with a patient's ability to sign informed consent, cooperate and participate in the study, or interfere with the interpretation of the results.
* History of allogeneic transplant
* Known HIV or Hepatitis B or C (active, previously treated or both)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2008-10; Primary Completion 2009-08 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amelia Zelnak, MD, Principal Investigator — Emory University Winship Cancer Institute
Locations (1):
- Emory University Winship Cancer Institute, Atlanta, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Arm Study: All patients enrolled on clinical trial will receive gemcitabine and oxaliplatin.
Period: Overall Study
Arm/Group | Single Arm Study
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm Study
Number analyzed (Participants) | 6
Age Continuous [Median (Full Range); unit: participants] | 55 [32 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Complete Response, Partial Response, Progressive Disease and Stable Disease.
Description: A sum of the longest diameter(LD) for all target lesions will be calculated and reported as the baseline sum LD.
  Complete Response (CR): Disappearance of all target lesions Partial Response (PR): At least a 30% decrease in the sum of the LD of target lesions, taking as reference the baseline sum LD Progressive Disease (PD):At least a 20% increase in the sum of the LD of target lesions.
  Stable Disease (SD):Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started.
Time Frame: 8 weeks
Measure: Number; unit: participants
Arm/Group | Gemcitabine and Oxaliplatin
Number analyzed (Participants) | 6
participants
  Stable Disease | 4
  Partial Response | 2

2. Secondary Outcome: Overall Survival From Time of Study Entry
Description: The number of weeks patient survived from the time of patient entry. The time frame reflects the time the first patient was entered into the study to the time till the last patient survived.
  Note: Not all patients started the study at the same time so the time frame is different from the full range.
  The full range reflects the least number of weeks a patient survived to the most number of weeks a patient survived.
Time Frame: 132 weeks
Measure: Median (Full Range); unit: Weeks
Arm/Group | Gemcitabine and Oxaliplatin
Number analyzed (Participants) | 6
Weeks | 62 [13 to 86]

ADVERSE EVENTS:
Arm/Group | Single Arm Study
Serious Adverse Events (participants affected / at risk) | 2/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm Study (N=6)
Infection (Infections and infestations) | 1 (6)
Neutropenia (Blood and lymphatic system disorders) | 1 (6)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single Arm Study (N=6)
Platelets (Blood and lymphatic system disorders) | 2
Hemoglobin (Blood and lymphatic system disorders) | 1
Neuropathy (Nervous system disorders) | 1
Fatigue (General disorders) | 1
Nausea (General disorders) | 2

LIMITATIONS AND CAVEATS:
Early termination of the study due to slow accrual

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes